CLINICAL TRIAL: NCT07184632
Title: A Study Investigating Safety, Tolerability and Efficacy of Once-weekly NNC0662-0419 in Participants Living With Overweight or Obesity
Brief Title: A Research Study on How Well Different Doses of the Medicine NNC0662-0419 Help People Living With Overweight or Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9662-8110; U1111-1317-2736 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0662-0419 (Experimental): Participants will be randomized to receive NNC0662-0419 subcutaneously (s.c.). The study will be conducted in 3 parts. Part A: Multiple ascending dose (MAD), Part B: Dose range finding (DFR) and Part C (2-week escalation).
  Interventions: Drug: NNC0662-0419
- Placebo (Placebo Comparator): Participant will be randomized to receive placebo in:
  The study will be conducted in 3 parts. Part A: Multiple ascending dose (MAD), Part B: Dose range finding (DFR) and Part C (2-week escalation).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0662-0419 — NNC0662-0419 will be administered subcutaneously.
  Arms: NNC0662-0419
Drug: Placebo — Placebo matched to NNC0662-0419 will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
This study tests how well different doses of the medicine NNC0662-0419 help people living with overweight or obesity. The purpose of the study is to find out if NNC0662-0419 is safe and effective for treating people living with overweight or obesity. There are 2 study treatments in this study, participants will get either NNC0662-0419, the treatment being tested or placebo, a treatment that has no active medicine in it. NNC0662-0419 is a new medicine which cannot be pre-scribed by doctors but has previously been tested in humans.

ELIGIBILITY:
Inclusion criteria

* Male or female (sex at birth).
* Age at the time of signing the informed consent:

  * For Part A:18-55 years (both inclusive)
  * For Part B and Part C: 18-65 years (both inclusive)
* Body Mass Index (BMI) at screening (overweight should be due to excess adipose tissue, as judged by the investigator):

  * For Part A: 27.0-39.9 kilogram per square meter(kg/m^2) (both inclusive)
  * For Part B and Part C:

    1. Greater than or equal to (≥) 27.0 kg/m^2 with the presence of at least one weight-related comorbidity (e.g. hypertension, dyslipidaemia, obstructive sleep apnoea or CV disease), or
    2. Greater than or equal to (≥) 30.0 kg/m^2
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as-judged by the investigator.
* Willingness to obtain a high weight loss (greater than [>] 25 percent [%]).

Exclusion criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Treatment with any compound containing Glucagon-Like Peptide 1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP) or amylin receptor agonism within 90 days before screening.
* Any condition, unwillingness or inability, which in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
* 2nd or 3rd degree atrioventricular-block, prolongation of the QRS complex over 120 millisecond (ms), or of the corrected QT interval by Fridericia (QTcF) calculation over 450 ms (females) or 430 ms (males), or any other clinically significant abnormal ECG results as judged by the investigator, at screening.
* Glycosylated haemoglobin (HbA1c) greater than or equal to (≥) 6.5% (48 millimoles per mole [mmol/mol]) at screening.
* History of type 1 or type 2 diabetes mellitus.
* Calcitonin greater than or equal to (≥) 50 nanogram per litre (ng/L) at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of treatment-emergent adverse events (TEAE) | From baseline (week 0) to end of study (up to week 44)
  Measured as number of events.
Part B: Relative change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured as percentage (%).
Part C: Occurrence of premature treatment discontinuation (Yes/No) | At end of treatment (week 24)
  Measured as count of participants.

SECONDARY OUTCOMES:
Part A: Relative change in body weight | From baseline (week 0) to end of treatment (up to week 40)
  Measured as percentage (%).
Part A: Change in body weight | From baseline (week 0) to end of treatment (up to week 40)
  Measured in kilograms (kg).
Part A: AUC; the area under the NNC0662-0419 plasma concentration-time curve | From pre-dose on day 1 to completion of the end of study visit (up to week 44)
  Measured in hours*nanomole per litre (h*nmol/L).
Part A: Cmax; the maximum plasma concentration of NNC0662-0419 | From pre-dose on day 1 to completion of the end of study visit (up to week 44)
  Measured in nanomole per litre (nmol/L).
Part B: Change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured in kg.
Part B: Body weight reduction greater than or equal to (≥) 5% (Yes/No) | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Part B: Body weight reduction ≥ 10% (Yes/No) | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Part B: Body weight reduction ≥ 15% (Yes/No) | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Part B: Body weight reduction ≥ 20% (Yes/No) | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Part B: Body weight reduction ≥ 25% (Yes/No) | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Part B: Number of treatment emergent adverse events (TEAE) | From baseline (week 0) to end of study (week 39)
  Measured as number of events.
Part C: Number of treatment emergent adverse events (TEAE) | From baseline (week 0) to end of study (week 27)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Celerion, Phoenix, Tempe, Arizona
  - Celerion, Lincoln, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: https://novonordisk-trials.com